CLINICAL TRIAL: NCT01241513
Title: Modulation of Oxygen Sensor Reactivity to Mimic Altitude Acclimatization
Brief Title: Induced Changes in Ventilatory Responsiveness and Altitude Exposure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Results of preliminary analyses showed no reason to continue the study
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H10-13
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Effects of High Altitude; Hypoxia; Inadequate or Impaired Breathing Pattern or Ventilation; Abnormal Blood Oxygen Pressure
Keywords: glutathione; redox status; carotid body chemosensitivity; ventilation
MeSH Terms: conditions — Altitude Sickness; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetyl-L-Cysteine (Experimental): N-Acetyl-L-Cysteine
  Interventions: Drug: NAC
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAC — NAC provided to determine if beneficial at altitude
  Other Names: NAC Accy
  Arms: N-acetyl-L-Cysteine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine if a drug (acetyl-cysteine or ACCY) can increase the amount of oxygen in your body at a high altitude of 11,500 feet. ACCY is approved by the Food and Drug Administration (FDA) as a treatment or antidote for Tylenol overdoses. Other forms of ACCY are also sold over-the-counter as nutritional supplements. In this study, the FDA-approved form of ACCY will be used "off-label" (meaning in a way not approved by the FDA).

This study is being conducted by researchers from the United States Army Research Institute of Environmental Medicine (USARIEM). The study will take place in the Altitude Chamber located in the basement of USARIEM. A total of approximately 30 volunteers (men and women, military and civilians) will take part in the study. They can expect to be in the study for a minimum of a few hours each day for two weeks.

The investigators hypothesize that ACCY will improve ventilation and oxygenation while at altitude.

DETAILED DESCRIPTION:
This study will determine if modulating reduction/oxidation (redox) status through a temporary increase in the blood ratio of reduced-to-oxidized glutathione (i.e., GSH/GSSG) will increase carotid body chemosensitivity and thus increase ventilation and arterial oxygen saturation (SaO2) during 32 hours of hypobaric hypoxia exposure to 3500 m (11,500 feet). To that end, the study will use an FDA-approved oral suspension form of acetylcysteine (ACCY) to modulate blood redox status under controlled conditions in the Hypobaric Chamber Facility at the USARIEM. Up to 30 healthy, active-duty military personnel or civilians from the local area will be recruited. Two independent treatment groups (placebo and ACCY; up to 15 in each group) will be assessed at sea level and altitude using a between-group experimental design. The two groups will be matched as closely as possible by age, ventilation, fitness, and gender prior to treatment assignment. Neither the staff nor the volunteers will know the treatment received by the groups until the study is completed. Included will be only those men and women who: are 18 to 39 years old, were born at altitudes below 2100 m (7000 feet), are not taking medications that interfere with oxygen delivery and transport (includes sedatives, sleeping aids, tranquilizers and any medication that depresses ventilation, diuretics, alpha and beta blockers); and have no evidence of any physical, mental, and/or medical conditions that would make the proposed study relatively more hazardous. All volunteers will participate over the two-week long study period in multiple standardized assessments that include resting (e.g., resting ventilation, SaO2, questionnaires), sleeping (e.g., heart rate, SaO2) and exercise (e.g., steady-state and time-trial performance, SaO2) measurements. The potential risks to test volunteers include the risks associated with hypobaric hypoxia exposure (e.g., acute mountain sickness [AMS; headache, nausea, insomnia]) and those associated with exercise (e.g., acute musculoskeletal strains and sprains, blisters). The investigators are not aware of any studies reporting problems during oral administration of ACCY in the doses or duration to be used in the present study. There are no direct benefits to the volunteers, except the knowledge of how well they performed at altitude and on the tests in which they participated. If the use of ACCY proves effective at altitude, then soldiers deployed to altitude in the future may have a means to beneficially increase ventilation and SaO2 in a manner similar to that experienced during natural altitude acclimatization.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Volunteers with the following criteria will be EXCLUDED from participation:

Less than 18 years of age Greater than 39 years of age Born at altitudes greater than 2134 m (7000 ft) Living in areas that are more than 1220 m (4,000 feet), or have traveled to areas that are more than 1220 m for more than a few days within the last 2 months.

Abnormal [Hb]/Hct levels or presence of hemoglobin S Known allergies to sulfonamide derivatives Smokers who smoke more than 5 cigarettes per day Tobacco chewers If military, unable to pass the 2-mi run portion of the Army Physical Fitness Test, or equivalent If civilian, not currently running or exercising for at least 20 min/day, 3X/week in "aerobic" activities (e.g., running, biking. swimming, basketball, etc) If they do not want to walk or run multiple times for 1 to 3 hours on a treadmill Unable to meet the U.S. Army height/weight standards Not willing to sleep in bunk beds in a small room (8 feet by 8 feet) with 1 to 3 other volunteers (male and/or female) for 3 nights. If they are claustrophobic Women who are pregnant or planning to conceive during the study period Women who are not willing to take urine pregnancy tests Not willing to drink an eight ounce solution of diet soda that may contain ACCY up to three times per day and then not willing to suck on a peppermint mint right after drinking the solution.

Taking medications that interfere with oxygen delivery and transport (Includes sedatives, sleeping aids, tranquilizers and any medication that depresses ventilation, diuretics, alpha and beta blockers) Evidence of any physical, mental, and/or medical conditions that would make the proposed studies relatively more hazardous. Evidence of prior HAPE or HACE diagnosis Evidence of apnea or other sleeping disorders Evidence of asthma If applicable, unwilling to stop taking all supplements for the two weeks of participation If applicable, all medications (prescription or over-the-counter) must be approved by the PI, and/or the OMSO.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2013-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Fulco, ScD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants withdrew prior to any testing
Groups:
- N-acetylcysteine: Active drug group
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started | 10 | 9
Completed | 10 (Study has been completed) | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- N-acetylcysteine (NAC): NAC
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine (NAC) | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (3) | 22 (3) | 22 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Arterial Oxygen Saturation
Description: Finger Pulse Oximetry to measure arterial oxygen saturation
Time Frame: Day 4 of treatment during acute altitude exposure
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Placebo Group: Placebo (Diet soda only)
- NAC Group: N-acetyl-L-Cysteine (800 mg T.I.D. in diet soda) for 4 days
Arm/Group | Placebo Group | NAC Group
Number analyzed (Participants) | 9 | 10
percentage of oxygen saturation | 82 (10) | 79 (12)

ADVERSE EVENTS:
Description: Adverse events can not be reported by intervention group because the data were not unblinded for data analyse. Based on results of preliminary analyses, the blind was not broken to further parse out the data for adverse events.
Arm/Group | NAC Group and Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 6/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC Group and Placebo Group (N=19)
Delayed patella tendon soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — recovered, finished study
back soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — aggravation of previously undisclosed condition
foot soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — expected post exercise
nausea and vomiting (Gastrointestinal disorders) | 1 (2) — determined to be due to caffeine withdrawal
acute mountain sickness (General disorders) | 1 (1) — expected adverse event; subject ended altitude exposure 4 hours early
knee injury (Musculoskeletal and connective tissue disorders) | 1 (1) — not study related

LIMITATIONS AND CAVEATS:
Study terminated due to results of preliminary analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No